CLINICAL TRIAL: NCT06213064
Title: A Direct-to-Consumer, Randomized, Double-blind, Placebo-controlled, Double Cross-over Study Investigating the Effect of Specific Cannabinoid Products on Motivation, Energy Level, Focus, and Appetite in Healthy Adults
Brief Title: A Direct-to-Consumer Study Investigating the Effect of Specific Cannabinoid Products on Motivation, Energy Level, Focus, and Appetite in Healthy Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Phylos Bioscience, Inc. (Industry)
Collaborators: People Science, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PS04
Record Dates: First submitted 2023-11-14; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Motivation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Product, THC Only Product, Placebo: All study participants will receive and cross-over into each group: study product, thc-only product, and placebo groups.
  Study Product Ingredient List:
  Active Ingredients: 10mg THCV, 5mg THC Tapioca syrup, sugar, water, pectin, citric acid, natural flavors*, coconut oil, sodium citrate, cannabis extract, soy lecithin,
  Infused THC Gummy Ingredient List:
  Active Ingredients: 5mg THC Tapioca syrup, sugar, water, pectin, citric acid, natural flavors*, coconut oil, sodium citrate, cannabis extract, soy lecithin, THC.
  Non-infused Placebo Gummy Ingredient List:
  Tapioca syrup, sugar, water, pectin, citric acid, natural flavors*, coconut oil, sodium citrate, soy lecithin.
  Interventions: Behavioral: Study Product, THC Product, Placebo

INTERVENTIONS:
Behavioral: Study Product, THC Product, Placebo — Participants will complete up to a seven week study consisting of screening period, baseline period, up to a 21-day product use period with a total of 9 product use sessions. Screening assessments, baseline questions, product use period questionnaires, adverse event reporting, and end of study experience survey data will be collected. This study will be conducted remotely and will use a web-based data collection platform, Consumer Health Learning and Organizing Ecosystem (Chloe), by People Science where participants will complete study assessments using the Chloe app during the course of the study. Participants will receive the study product during the baseline period. Demographic and medical history data will be collected for the study.

SUMMARY:
Tetrahydrocannabivarin (THCV) is a rare cannabinoid and is a homologue of THC that differs only in the length of the alkyl side chain (3C vs 5C, respectively). Pre-clinical and clinical trials have shown that THCV has medical potential as a neuroprotectant, anti-inflammatory, anti-anxiety, and most notably as a therapeutic to improve glycemic control in type 2 diabetic patients.

Several THCV products are available in states with recreational cannabis. Anecdotal reports from adult cannabis users indicate that THCV provides an energizing, focusing and euphoric high-while still creating a lucid, uplifting experience. Additionally, unlike THC-dominant products, THCV was not reported to increase appetite. Other anecdotal comments referring to increased ability to focus for long periods of time and being more active were common.

Given anecdotal evidence, which shows that THCV is activating and improving focus, this provides rationale and justification to conduct a clinical research study to further test and understand whether THCV improves motivation, focus, level of energy, and does not stimulate appetite in healthy adults.

DETAILED DESCRIPTION:
The rationale for this study is to determine the effect of a consumer-grade, state-legal formulation of cannabinoids including Tetrahydrocannabivarin (THCV) on motivation, energy level, focus, and appetite. A consumer-driven, decentralized observational clinical research study is therefore well suited to examine the effect of this formulation in healthy individuals.

The investigators will examine the outcomes in a broad age-range of adults who have chosen to try these products. The study will incorporate participant reported outcomes and surveys collected after each product use session to engage the participant in their typical day-to-day activities. There is no "physician-patient" relationship as part of this research since the participant as a consumer is making the informed choice to take the products and take part in the observational process with self-reported measures. Findings from this study will contribute knowledge toward the design of future cannabis research studies and the improvement of the product formulation.

A new study questionnaire was developed as no existing questionnaire would be able to capture all interest areas of this study in a holistic manner. Other questionnaires related to focus, attention, concentration, fatigue, work, and motivation were assessed and used to support the study questionnaire development.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults age > 21 years old
2. Work / study / play in an environment that requires focus
3. Able to read and understand English
4. Able to read, understand, and provide informed consent
5. Able to use a personal smartphone device and download Chloe by People Science
6. Able to complete study assessments over the course of up to 14 days
7. Familiar with the use of cannabis and its effects
8. Able to tolerate at least 5mg THC
9. Willingness to abstain from use of any THC containing products during study product use days
10. Willingness to abstain from use of alcohol during study product use days
11. Greater Los Angeles area residents only

Exclusion Criteria:

1. Participants who do not have a smartphone and/or internet access
2. Any known adverse effects from taking cannabis
3. Concomitant Therapies: Currently taking medication for ADHD or psychotropic medications
4. Other Illnesses or Conditions: Participants who have the following co-morbidities are excluded:

   1. History or currently undergoing product use for substance abuse disorders
   2. Currently pregnant, planning to become pregnant within the next month, or breastfeeding
   3. Allergies to formulation ingredients
   4. Current or prior psychotic disorder
   5. Immunosuppressive product uses, including organ transplant participants, active immunotherapy for cancer product use
   6. Any condition that is considered by investigator to be a contraindication to cannabis (e.g. specific drug-use interaction, unstable cardiac arrhythmia)

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample size for this study will be approximately 58 healthy volunteers who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
To observe the effect of various cannabinoid-containing products on motivation. | 3 weeks
  Change in average motivation score by 1 point as measured by a 10-point visual analogue rating scale (VAS) collected between cannabinoid and placebo use sessions. The scale is between 1-10, where 1 denotes 'Strongly Disagree' and 10 denotes 'Strongly Agree.'

SECONDARY OUTCOMES:
To observe the effect of cannabinoid products on motivation, energy level, focus, and appetite (MEFA). | 3 weeks
  Change in average score by 1 point as measured by a 10-point visual analogue rating scale (VAS) between the cannabinoid and placebo use sessions. The scale is between 1-10, where 1 denotes 'Strongly Disagree' and 10 denotes 'Strongly Agree.'

OTHER OUTCOMES:
To observe changes in overall symptoms and quality of life. | 3 weeks
  Changes in overall symptoms and quality of life to be assessed based on a qualitative evaluation of study participant experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Craft, MD, Principal Investigator — People Science, Inc.
Locations (1):
- People Science, Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data is there own. Participant consent will need to be obtained for other researchers.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT06213064/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT06213064/ICF_001.pdf